CLINICAL TRIAL: NCT00571324
Title: An Open Label Pilot Study of the Effects of the Glucagon-like Peptide-1 Receptor Antagonist, Exendin-(9-39) on Glycemic Control in Subjects With Congenital Hyperinsulinism
Brief Title: Effect of Exendin-(9-39) on Glycemic Control in Subjects With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diva De Leon (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Diva De Leon, M.D. Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2007-1-5131; R03DK078535-01 (NIH)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Congenital Hyperinsulinism
Keywords: hyperinsulinism; hypoglycemia; KATP channel; Kir6.2
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism; Hypoglycemia | interventions — exendin (9-39)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exendin-(9-39) first, the Vehicle (Experimental): Exendin-(9-39) will be administered intravenously (IV) after an overnight fast. Exendin-(9-39) will be infused over 6 hours with the dose slowly escalating from 100pmol/kg/min for 2 hours, then 300pmol/kg/min for another 2 hours followed by 500pmol/kg/min for the last 2 hours of the infusion. The following day, after another overnight fast, normal saline (control) vehicle infusion will be administered intravenously (IV) over 6 hours. During both infusions, blood glucose levels will be measured every 20 minutes.
  Interventions: Drug: Exendin-(9-39); Other: Vehicle
- Vehicle first, then Exendin-(9-39) (Placebo Comparator): Normal saline vehicle infusion will be administered intravenously (IV) after an overnight fast. The infusion will be given over 6 hours. The following day, after another overnight fast, Exendin-(9-39) will be infused over 6 hours with the dose slowly escalating from 100pmol/kg/min for 2 hours, then 300pmol/kg/min for another 2 hours followed by 500pmol/kg/min for the last 2 hours of the infusion. During both infusions, blood glucose levels will be measured every 20 minutes.
  Interventions: Drug: Exendin-(9-39); Other: Vehicle

INTERVENTIONS:
Drug: Exendin-(9-39) — A short term intravenous infusion of the study drug, exendin-(9-39), will be given over 6 hours.
Other: Vehicle — A short term intravenous infusion of normal saline, or the vehicle, will be given over 6 hours.
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine if Exendin-(9-39), an antagonist of the glucagon-like peptide-1 (GLP-1) receptor with effects on the pancreatic beta cell, increases fasting blood glucose levels in subjects with congenital hyperinsulinism.

DETAILED DESCRIPTION:
This is an open-label, pilot study , to determine if Exendin-(9-39), an antagonist of the glucagon-like peptide-1 (GLP-1) receptor with effects on the pancreatic beta cells, increases fasting blood glucose levels in subjects with congenital hyperinsulinism. Our overall hypothesis is that abnormal GLP-1 secretion resulting from dysfunctional nutrient sensing in intestinal L-cells plays a role in the dysregulated insulin secretion characteristic of this disorder, and that antagonism of the GLP-1 receptor will increase fasting blood glucose levels.

Aim 1. To evaluate the dose of exendin-(9-39) required to elevate fasting blood glucose levels in subjects with congenital hyperinsulinism due to KATP channel mutations.

Aim 2. To determine therapeutic plasma levels, plasma half-life and pharmacokinetics of exendin-(9-39) during an intravenous short-term infusion in subjects with congenital hyperinsulinism due to Adenosine triphosphate (ATP)-sensitive potassium channel (KATP) mutations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with congenital hyperinsulinism

Exclusion Criteria:

* Acute medical illness
* History of other systemic chronic disease such as cardiac failure, renal insufficiency, hepatic insufficiency, chronic obstructive pulmonary disease, anemia, or uncontrolled hypertension
* Pregnancy
* Diabetes mellitus
* Use of medications that affect glucose metabolism, such as glucocorticoids, beta agonists, diazoxide and octreotide.
* Subjects will be eligible to participate 48 hrs after the last dose of octreotide and 72 hrs after last dose of diazoxide

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diva D De Leon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Calabria AC, Li C, Gallagher PR, Stanley CA, De Leon DD. GLP-1 receptor antagonist exendin-(9-39) elevates fasting blood glucose levels in congenital hyperinsulinism owing to inactivating mutations in the ATP-sensitive K+ channel. Diabetes. 2012 Oct;61(10):2585-91. doi: 10.2337/db12-0166. Epub 2012 Aug 1. PMID 22855730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with confirmed genetic and clinical diagnosis of Adenosine triphosphate (ATP)-sensitive potassium channels (KATP) hyperinsulinism were recruited from the Hyperinsulinism Center at the Children's Hospital of Philadelphia
Groups:
- Exendin-(9-39) First, the Vehicle: Exendin-(9-39) was administered intravenously (IV) after an overnight fast. Exendin-(9-39) was infused over 6 hours with the dose slowly escalating from 100pmol/kg/min for 2 hours, then 300pmol/kg/min for another 2 hours followed by 500pmol/kg/min for the last 2 hours of the infusion. The following day, after another overnight fast, normal saline (control) vehicle infusion was administered intravenously (IV) over 6 hours. During both infusions, blood glucose levels were measured every 20 minutes.
- Vehicle First, Then Exendin-(9-39): Normal saline vehicle infusion was administered intravenously (IV) after an overnight fast. The infusion was given over 6 hours. The following day, after another overnight fast, Exendin-(9-39) was infused over 6 hours with the dose slowly escalating from 100pmol/kg/min for 2 hours, then 300pmol/kg/min for another 2 hours followed by 500pmol/kg/min for the last 2 hours of the infusion. During both infusions, blood glucose levels were measured every 20 minutes.
Period: Intervention 1 (7 Hours)
Arm/Group | Exendin-(9-39) First, the Vehicle | Vehicle First, Then Exendin-(9-39)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Intervention 2 (7 Hours)
Arm/Group | Exendin-(9-39) First, the Vehicle | Vehicle First, Then Exendin-(9-39)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subject Population: All subjects enrolled and treated in the protocol served as their own control. Because of this and the small sample size, baseline characteristic data is presented together.
Arm/Group | Subject Population
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Mutation (ABCC8) [Number; unit: participants]
  Heterozygous dominant ABCC8 mutations | 6
  Homozygous common recessive Ashkenazi mutation | 2
  Compound heterozygous recessive ABCC8 mutations | 1
Pancreatectomy [Number; unit: participants] — Whether subject has undergone prior pancreatectomy during infancy and if so, what percent of the pancreas was removed.
  participants
    None | 6
    85% Pancreatectomy | 1
    95% Pancreatectomy | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose Area Under the Curve (AUC 0-6h)
Description: To examine the effect of Exendin-(9-39) on fasting blood glucose levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (Time 0), and then every 20 minutes until 6 hours after the start of the infusion. Using this information, the mean blood glucose area under the curve (AUC) from the start of the infusion to the end of the infusion (360 minutes) was calculated for each both Exendin-(9-39) and vehicle and compared.
Time Frame: 6 hours
Population: Subjects served as their own control for comparison between effects of Exendin-(9-39) and the normal saline vehicle.
Measure: Mean (Standard Error); unit: mmol*min/L
Groups:
- Exendin-(9-39): Exendin-(9-39) was administered intravenously (IV) after an overnight fast. Exendin-(9-39) was infused over 6 hours with the dose slowly escalating from 100pmol/kg/min for 2 hours, then 300pmol/kg/min for another 2 hours followed by 500pmol/kg/min for the last 2 hours of the infusion.
- Vehicle: Normal saline vehicle infusion was administered intravenously (IV) after an overnight fast. The infusion was given over 6 hours.
Arm/Group | Exendin-(9-39) | Vehicle
Number analyzed (Participants) | 9 | 9
mmol*min/L | 2,096 (454) | 1,678 (281)

2. Secondary Outcome: Mean Plasma Insulin Area Under the Curve (AUC 0-6h)
Description: To examine the effect of Exendin-(9-39) on plasma insulin levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (Time 0), and then every 20 minutes until 6 hours after the start of the infusion. Using this information, the mean plasma insulin area under the curve (AUC) from the start of the infusion to the end of the infusion (360 minutes) was calculated for each both Exendin-(9-39) and vehicle and compared.
Time Frame: 6 hours
Population: Subjects served as their own control for comparison between effects of Exendin-(9-39) and the normal saline vehicle.
Measure: Mean (Standard Error); unit: pmol*min/L
Arm/Group | Exendin-(9-39) | Vehicle
Number analyzed (Participants) | 9 | 9
pmol*min/L | 21,016 (7,410) | 25,842 (12,397)

3. Secondary Outcome: Mean Plasma Glucagon Area Under the Curve (AUC 0-6h)
Description: To examine the effect of Exendin-(9-39) on plasma glucagon levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (Time 0), and then every 20 minutes until 6 hours after the start of the infusion. Using this information, the mean plasma glucagon area under the curve (AUC) from the start of the infusion to the end of the infusion (360 minutes) was calculated for each both Exendin-(9-39) and vehicle and compared.
Time Frame: 6 hours
Population: Subjects served as their own control for comparison between effects of Exendin-(9-39) and the normal saline vehicle.
Measure: Mean (Standard Error); unit: pg*min/dL
Arm/Group | Exendin-(9-39) | Vehicle
Number analyzed (Participants) | 9 | 9
pg*min/dL | 21,243 (5,836) | 21,867 (4,432)

4. Secondary Outcome: Mean Plasma Intact Glucagon-Like Peptide-1 (GLP-1) Area Under the Curve (AUC 0-6h)
Description: To examine the effect of Exendin-(9-39) on plasma intact glucagon-like Peptide-1 (GLP-1) levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (Time 0), and then every 20 minutes until 6 hours after the start of the infusion. Using this information, the mean intact GLP-1 area under the curve (AUC) from the start of the infusion to the end of the infusion (360 minutes) was calculated for each both Exendin-(9-39) and vehicle and compared.
Time Frame: 6 hours
Population: Subjects served as their own control for comparison between effects of Exendin-(9-39) and the normal saline vehicle.
Measure: Mean (Standard Error); unit: pmol*min/L
Arm/Group | Exendin-(9-39) | Vehicle
Number analyzed (Participants) | 9 | 9
pmol*min/L | 1,970 (1,284) | 1,992 (1,203)

ADVERSE EVENTS:
Time Frame: 30 days following the last administration of study treatment (either Exendin-(9-39) or vehicle)
Arm/Group | Exendin-(9-39) | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exendin-(9-39) (N=9) | Vehicle (N=9)
Hypoglycemia (Endocrine disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to safety concerns subjects with symptomatic hypoglycemia were rescued with dextrose to maintain glucose levels >60mg/dL limiting detectable treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes